CLINICAL TRIAL: NCT00642421
Title: Safety and Biological Activity of a New Prolonged Release Formulation of Octreotide Acetate, C2l-OCT-01 PR, Administered Intra Muscularly Every 4, 5 or 6 Weeks in Acromegalic Patients
Brief Title: Safety and Biological Activity of C2L-OCT-01 PR in Acromegalic Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Commercial reasons
Sponsor: Ambrilia Biopharma, Inc. (Industry)
Responsible Party: Bonabes de Rouge, M.D./Senior Executive Vice-President & Chief Scientist Officer, Ambrilia Biopharma, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C2L-OCT-01 PR-303
Record Dates: First submitted 2008-03-21; First posted 2008-03-25 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2010-02

CONDITIONS: Acromegaly
Keywords: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Population A (Experimental): Based on the dose of their previous Sandostatin-LAR treatment, Population A will receive 10 or 20 mg of C2L-OCT-01 PR at 5-week intervals.
  Interventions: Drug: C2L-OCT-01 PR, 10 or 20 mg
- Population B (Experimental): Population B, naive patients and patients who have stopped their treatment with prolonged release octreotide for at least 12 weeks, will receive 20 mg C2L-OCT-01 PR at 5-week intervals.
  Interventions: Drug: C2L-OCT-01 PR, 20 mg

INTERVENTIONS:
Drug: C2L-OCT-01 PR, 10 or 20 mg — The first three injections of study medication will be given at V1 (Day 1), V2 (35 days) and V3 (70 days). Dose titration and/or injection interval adjustment will be allowed during the Treatment Period should any patients have a mean GH concentration below 1.0 ng/mL or above 2.5 ng/mL. Dose titration (10, 20 or 30 mg) and/or injection interval adjustment (4, 5 or 6 weeks) will be allowed at V3, V6 and V9 based on clinical symptoms and the mean GH concentration determined at V2, V5 and V8.
  Other Names: octreotide acetate
  Arms: Population A
Drug: C2L-OCT-01 PR, 20 mg — The first three injections of study medication will be given at V1 (Day 1), V2 (Day 35) and V3 (Day 70). Dose titration and/or injection interval adjustment will be allowed during the Treatment Period should any patients have a mean GH concentration below 1.0 ng/mL or above 2.5 ng/mL. Dose titration (10, 20 or 30 mg) and/or injection interval adjustment (4, 5 or 6 weeks) will be allowed at V3, V6 and V9 based on clinical symptoms and the mean GH concentration determined at V2, V5 and V8.
  Other Names: octreotide acetate
  Arms: Population B

SUMMARY:
The purpose of this study is to assess the safety profile of a new prolonged release formulation of octreotide acetate, C2L-OCT-01 PR, administered intra muscularly every 4, 5 or 6 weeks in acromegalic patients.

ELIGIBILITY:
To be eligible for entry in this study, patient must:

* Be greater than or equal to 18 years of age.
* Have a confirmed diagnosis of acromegaly based on the following criteria:

  1. Typical clinical features and
  2. Mean GH concentration > 1.0 ng/mL following an oral glucose tolerance test (OGTT) and
  3. Elevated serum IGF-1 levels above gender- and age- matched values.
* Fall into one of the following categories:

  1. Has been treated for at least the last 12 weeks with Sandostatin LAR® 10 mg or 20 mg, every 28 days with well-controlled symptoms of acromegaly and GH concentration < 2.5 ng/mL at screening or
  2. Be naïve to prolonged release octreotide with a demonstrated tolerance response to a 7-day administration of Sandostatin® immediate release (50 µg s.c. t.i.d.) or
  3. If previously treated with prolonged release octreotide, has stopped such treatment for at least 12 weeks prior to screening.
* If female and of childbearing potential, must have a negative pregnancy test at screening and be using adequate means of birth control (i.e., oral or trans-dermal contraceptive drugs, intra-uterine device, diaphragm) during the study.
* Have the ability to understand the requirements of the study, provide written informed consent to participate in this study and agree to abide by the study restrictions.

Exclusion Criteria

To be eligible for entry in this study, patient must NOT:

* If female, be pregnant or lactating.
* Have been treated with a GH receptor antagonist (pegvisomant) within the last 12 weeks.
* Have used a dopamine agonist within the last 30 days.
* Have undergone pituitary surgery within the last 12 weeks.
* Have undergone radiotherapy within the last two years.
* Have any contraindication (hypersensitivity to octreotide formulation) or non-responders to Sandostatin-LAR® treatment.
* Be currently treated with Sandostatin-LAR® and have symptoms of acromegaly that would justify, in the Investigator's opinion, a dose modification.
* Be receiving Sandostatin-LAR® administration every < 21 or > 35 days.
* Have a liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis, or has persistent ALT, AST > 2 X ULN, serum creatinine > 2 X ULN, serum bilirubin > 2 X ULN.
* Have any other conditions that could result in altered GH or IGF-1 levels (such as anorexia nervosa, Laron's syndrome, treatment with levodopa or narcotics analgesics, heroin abuse.)
* Have type I diabetes (insulin-dependent) or uncontrolled type II diabetes (non-insulin-dependent) as indicated by the presence of ketoacidosis or HbA1C greater than or equal to 10%.
* Have clinically significant signs and symptoms potentially related to a tumor compression of the optical chiasm, based on judgment of the investigator.
* Have symptomatic cholelithiasis.
* Have received an investigational drug or participated in a clinical trial within the last 30 days.
* Have clinically serious and/or unstable intercurrent infection, medical illnesses or conditions that are uncontrolled or whose control, in the opinion of the Investigator, may be jeopardized by participation in this study or by the complications of this therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
To assess the safety profile of a new prolonged release formulation of octreotide acetate, C2L-OCT-01 PR, administered intra muscularly every 4, 5 or 6 weeks in acromegalic patients. | 28-day screening period followed by a 48 to 52 week treatment period and concluding with a end of study visit at 56, 57 or 58 weeks.

SECONDARY OUTCOMES:
To assess biological and clinical activity of C2L-OCT-01 PR by examining the percentage of patients with mean growth hormone (GH) <2.5 ng/ml. | Screening, Visits 1 through 11, and End of Study Visit.
To assess the biologic and clinical activity of C2L-OCT-01 PR by examining the mean changes from baseline in GH and IGF-1 concentrations. | Screening, Visits 1 through 11, and End of Study Visit.
To assess the biologic and clinical activity of C2L-OCT-01 PR by examining the acromegaly severity index and patient's health status scores. | Screening, Visit 1 through 11, and End of Study Visit.
To assess biological and clinical activity of C2L-OCT-01 PR by examining the pituitary tumor size. | Screening, Visit 6 and End of Study Visit.

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Naudin, M.D., Study Director — Ambrilia Biopharma, Inc.
Locations (10):
- United States (5):
  - UCLA Medical Center Division of Neurosurgery, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - Kaleida Health/Diabetes Center of WNY, Buffalo, New York
  - The Cleveland Clinic, Cleveland, Ohio
  - VA Puget Sound Health Care System, Tacoma, Washington
- Republican Centre for Medical Rehabilitation and Water-therapy, Minsk, Belarus
- Semmelweis Egyetem Altalanos Orvostudomanyi, Budapest, Hungary
- Institute of Endocrinology "C.I. Parhon" Bucharest, Bucharest, Romania
- Institute of Endocrinology, University Clinical Center, Belgrade, Serbia
- V.P. Komisarenko Institute of Endocrinology and Metabolism, AMS Ukraine, Kiev, Ukraine